CLINICAL TRIAL: NCT02882022
Title: Evaluating Changes in Middle Ear Pressure Caused by CPAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to lack of participants
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bradley Kesser, MD, Associate professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19158
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Eustachian Tube Disorder
Keywords: Eustachian tube dysfunction; Audiometry
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPAP (Experimental): All participants will be included in this arm, and CPAP will be administered using a full face mask at incrementally increasing pressures. This will occur during a single session lasting no more than one hour.
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — A CPAP machine will be used to deliver positive pressure at various levels after which middle ear pressure and ear drums will be evaluated for changes.
  Other Names: CPAP

SUMMARY:
This study is an investigation into the effect that CPAP has on the pressure in the middle ear. It will evaluate the middle ear pressure and ear drum appearance at multiple levels of CPAP pressure delivered via a full face mask. These measurements will be used to determine optimal levels of CPAP to affect individual's middle ear pressure, particularly those with negative middle ear pressure due to Eustachian tube dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* No use of CPAP within past 30 days
* Individuals presenting to the UVA otolaryngology clinic who are otherwise healthy

Exclusion Criteria:

* Pre-existing cardiopulmonary disease that presents a risk with CPAP use
* Inability to tolerate CPAP
* Recent otologic surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Tympanometry | 1 minute
  Probes in the ear canal evaluate middle ear pressure

SECONDARY OUTCOMES:
Subjective sensation | 1 minute
  Patient reports if they felt their ears "pop"
Subjective symptom score | 1 minute
  A simple 7 question form regarding ear symptoms over the past month prior to trial involvement
Otoscopy | 1 minute
  An image of the ear drum is captured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Akbulut S, Demir MG, Salepci BM, Gungor GA, Demir N, Berk D, Cakan D. Efficacy of continuous positive airway pressure on middle ear atelectasis: A double-blind placebo-controlled clinical trial. Laryngoscope. 2016 Jul;126(7):1649-55. doi: 10.1002/lary.25735. Epub 2015 Oct 20. PMID 26485439
- [Background] Aksoy F, Yildirim YS, Ozturan O, Veyseller B, Cuhadaroglu C. Eustachian tube function in patients receiving continuous positive airway pressure treatment for sleep apnea syndrome. J Otolaryngol Head Neck Surg. 2010 Dec;39(6):752-6. PMID 21144374
- [Background] Drake-Lee AB, Casey WF, Ogg TW. Anaesthesia for myringotomy. The effect of nitrous oxide and intermittent positive pressure ventilation in children with secretory otitis media. Anaesthesia. 1983 Apr;38(4):314-8. doi: 10.1111/j.1365-2044.1983.tb10451.x. PMID 6342458
- [Background] Lin FY, Gurgel RK, Popelka GR, Capasso R. The effect of continuous positive airway pressure on middle ear pressure. Laryngoscope. 2012 Mar;122(3):688-90. doi: 10.1002/lary.22442. Epub 2012 Jan 17. PMID 22252535
- [Background] Sivri B, Sezen OS, Akbulut S, Coskuner T. The effect of continuous positive airway pressure on middle ear pressure. Laryngoscope. 2013 May;123(5):1300-4. doi: 10.1002/lary.23896. Epub 2013 Apr 2. PMID 23553241

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT02882022/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT02882022/ICF_001.pdf